CLINICAL TRIAL: NCT00897715
Title: Inflammation in CKD and CVD - The Role of Genetics and IL-1ra
Brief Title: Inflammation in Chronic Kidney Disease and Cardiovascular Disease - The Role of Genetics and Interleukin-1 Receptor Antagonist (IL-1ra)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDA-2-031-09S
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
Keywords: CKD; inflammation; CVD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Inflammation | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interleukin-1 receptor antagonist (Active Comparator): active drug
  Interventions: Drug: Rilonacept
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilonacept — 160 mg of rilonacept administered subcutaneously once a week for 12 weeks
  Other Names: Arcalyst
  Arms: Interleukin-1 receptor antagonist
Drug: Placebo — 160 mg of placebo administered subcutaneously once a week for 12 weeks
  Arms: Placebo

SUMMARY:
There has been an exponential growth in the number of people with Chronic Kidney Disease (CKD) needing dialysis or transplantation, increasing from 209,000 in 1991 to 472,000 in 2004. This is highly concerning due to both the human cost and the burden that it represents to the health care system. Recent comparison of the NHANES surveys showed that CKD prevalence increased from 10% in 1988-1994 to 13% in 1999-2004. Patients with CKD are more likely to die from premature cardiovascular death than to reach ESRD. In those that reach ESRD, cardiovascular disease (CVD) accounts for over half of the deaths in dialysis. The prevalence of CKD for the VA population is 20%, and 31.6% for diabetics, higher than in the general population. These observations emphasize the need of risk stratification, early detection, and prevention efforts with respect to CKD progression and the CVD burden that afflicts CKD through targeted interventions in high-risk groups (personalized medicine).

CKD is multifactorial, however familial aggregation of end-stage renal disease (ESRD) and CKD have been reported for all types of nephropathy underscoring "kidney disease genetic susceptibility ". Genetic predisposition to ESRD is stronger in African Africans. African Americans with a first-degree relative with ESRD have a 9-fold increase risk of ESRD vs. a 3-5 fold increase in whites.

Studies consistently show that CKD is an inflammatory process and that biomarkers of inflammation increase since early stages of CKD. CVD is also an inflammatory process, and genes that affect inflammation are associated with higher risk of CVD. Since inflammation is a common denominator of both disease processes (CKD and CVD), it is likely that genes that govern inflammation may be involved in both, the predisposition to CKD and the burden of CVD attributable to CKD. Additionally if inflammation plays a central role in the burden of CVD in CKD than drugs that modulate inflammation should impact both: CKD progression and non-traditional CV risk factors and CVD.

The overall goal of this proposal is to study genetic predisposition to CKD, and CVD risk in CKD through inflammatory pathways, and the effect that a potent anti-inflammatory intervention like interleukin 1 receptor antagonist (IL-1ra), will have in inflame patients with CKD stages 3&4. Specific Aims: 1) To determine if specific polymorphism/haplotypes, genotype combinations and gene-environmental interactions that can affect inflammation, available from the Third National Health and Nutrition Examination Survey (DNA data set), specifically in the CRP,IL-1, IL-10 and TNF- genes, are associated with CKD. 2) To determine if the specific polymorphisms and haplotypes studied in Aim 1 are associated with faster CKD progression and CV outcomes in a longitudinal cohort from the African American Study of Kidney Disease. 3)To determine if a targeted anti-inflammatory intervention, an IL-1 receptor antagonist, will modulate systemic inflammation, endothelial function, oxidative stress and urinary cytokines, the proposed surrogate markers of CVD and CKD progression in inflame patients with CKD stages 3&4.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* estimated glomerular filtration rate (eGFR) between 15-60 mL/min/1.73m2;
* Must be on stable regimens of medications that can affect inflammatory axis (Aspirin, Thiazolidinediones, statins);
* Willing and able to comply with clinic visits and study-related procedures;
* Provide signed informed consent.

Exclusion Criteria:

* Recent infection or hospitalization (within one month);
* History of active or chronic hepatitis B, history of active or chronic hepatitis C, human immunodeficiency virus (HIV), history of tuberculosis (patient must be purified protein derivate negative);
* Patients taking tumor necrosis factor (TNF) inhibitors, TNF blocker, interleukin-6 (IL-6) blockers or interleukin-1 (IL-1) blocking drugs;
* Patients on steroids or receiving any other immunosuppressive agent or anti-inflammatory drug (aspirin up to 325 mg a day is allowed) one month prior;
* Have clinically significant chronic lymphopenia (low white blood cell count);
* History of malignancy in the prior 5 years. Any history of melanoma or lymphoma;
* Life expectancy less than six months;
* Intolerance to the study medication;
* The use of any other investigational drug 30 days prior to enrollment or within five half-lives of the medication used;
* Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose;
* Currently receiving parenteral iron or scheduled to receive parenteral iron during the study;
* Uncontrolled diabetes mellitus (glycated hemoglobin > 10);
* high sensitivity c-reactive protein (hsCRP) <2mg/L or >30 mg/L;
* Body mass index (BMI) > 40;
* Known diagnosis of severe congestive heart failure with documented ejection fraction (EF) < 35%;
* Pregnant or breast-feeding women;
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

  * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2015-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Hung, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (2):
- United States (2):
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the VA Nashville between 01/2013 and 02/2015. Note that essentially the same study was also conducted at the University of Colorado (NCT01663103). Results were combined with Colorado for publication. However, the results reported here are only based on the subjects enrolled at the VA Nashville.
Pre-assignment Details: There is about a 2-week screening period between enrollment and assignment to a treatment group to access inclusion/exclusion criteria. Although 45 subjects were enrolled, only 15 subjects were assigned to a treatment group (30 subjects were screen failures).
Period: Overall Study
Arm/Group | Interleukin-1 Receptor Antagonist | Placebo
Started | 8 | 7
Completed | 6 | 6
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — increased risk of infection | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interleukin-1 Receptor Antagonist | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.5) | 67 (6.2) | 64 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in the Concentration of High Sensitivity C-Reactive Protein (hsCRP) From Baseline to 12 Weeks
Description: hsCRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation
Time Frame: baseline and 12 weeks
Population: The number of participants for analysis was based on those subjects who completed the 12-week study, as well as 2 subjects who withdrew but completed end-of-study procedures (1 in each group). The analysis was per protocol. Note that the results reported here are only based on the subjects enrolled at the VA Nashville.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Interleukin-1 Receptor Antagonist | Placebo
Number analyzed (Participants) | 7 | 7
mg/dl | -2.6 [-3.05 to -1.35] | 0.8 [-0.05 to 1.3]
Statistical Analysis 1: Comparison: Interleukin-1 Receptor Antagonist vs Placebo; For the primary specific aim, we will compare the mean percent change on hsCRP between the intervention arm and the placebo arm using linear regression. We anticipate that the intervention will conservatively decrease hsCRP by 54%; whereas, placebo will have no effect. Accordingly, we have estimated that we will need 24 subjects in the experimental arm and 24 controls to have an 80% power, with an alpha of 0.05 to detect the above mentioned effect size; Test type: Superiority or Other; p = 0.03, ANCOVA — 0.05 is the a priori threshold for statistical significance

2. Secondary Outcome: Change in Concentration of Interleukin-6 (IL-6) From Baseline to 12 Weeks
Description: IL-6 is a sensitive laboratory assay for serum levels of Interleukin-6, which is a pro-inflammatory cytokine that is used to evaluate the inflammatory response
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Interleukin-1 Receptor Antagonist | Placebo
Number analyzed (Participants) | 7 | 7
pg/ml | -0.63 [-0.98 to 0.00] | 0.05 [-0.18 to 0.53]
Statistical Analysis 1: Comparison: Interleukin-1 Receptor Antagonist vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA — 0.05 is the a priori threshold for statistical significance

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Interleukin-1 Receptor Antagonist | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 4/8 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interleukin-1 Receptor Antagonist (N=8) | Placebo (N=7)
back pain (General disorders) | 1 (2) | 0 (0)
injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nerve puncture (Nervous system disorders) | 0 (0) | 1 (1)
infection (Infections and infestations) | 0 (0) | 1 (1)
heart arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
burn (General disorders) | 1 (1) | 0 (0)
cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes